CLINICAL TRIAL: NCT04690400
Title: Adaptations From a Telehealth Stretching Exercise Program on Painful Conditions, Depression, Sleep and Functionality of Women With Fibromyalgia During the Covid-19 Pandemic: a Randomized Clinical Trial
Brief Title: Telehealth Stretching Exercise Program for Women With Fibromyalgia During the Covid-19 Pandemic
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Federal University of Pelotas (Other)
Responsible Party: Principal Investigator, Cristine Lima Alberton, PhD, Federal University of Pelotas
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 39305720.9.0000.5313
Record Dates: First submitted 2020-12-20; First posted 2020-12-30 (Actual); Last update posted 2021-12-30 (Actual); Status verified 2021-12

CONDITIONS: Fibromyalgia; Fibromyalgia, Primary
Keywords: Stretching exercise; Telehealth
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Intervention Model Description: This is a randomized, single-blinded, parallel, superiority, controlled trial. Participants, women with fibromyalgia, will be allocated to two groups, experimental and control, based on randomization sequence. Sequence will be generated by computer, with 1:1 ratio and blocks of random sizes that are not disclosed to ensure concealment. Allocation concealment will be implemented through a central randomization routine conducted by the same investigator that will generate the sequence. The allocation of participants will occur after the completion of baseline outcomes evaluations.
Who Masked: Outcomes Assessor
Masking Description: Blinding will be implemented for outcome assessor. The questionnaires and functional tests will be supervised remotely by an investigator blinded to the participant's group. Due to the type of interventions, the investigator conducting exercise sessions as well as participants are not blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active care group (Experimental): Participants will practice stretching exercises twice a week, at a distance and under the supervision of a professional, for 12 weeks. In addition, the experimental group will receive the same written guide and video of the comparator group.
  Interventions: Other: Experimental: Active care group
- Self-care group (Active Comparator): Participants will receive stretching advice by written guide and video with stretching exercises, to be performed individually, without distance supervision, for 12 weeks. Participants will be able to resolve questions about the protocol at any time, via telephone.
  Interventions: Other: Active Comparator: Self-care group

INTERVENTIONS:
Other: Experimental: Active care group — Stretching exercise program remotely supervised. Total of approximately 40 minutes per session by WhatsApp, individually and supervised by a professional (physiotherapist or physical education teacher). As recommended for flexibility improving, 30 seconds of stretching in each exercise will be perform fractionated (3 series of 10 seconds of static position at the point of moderate discomfort, with 10 seconds interval between series). There will be two stretching protocol models with exercises variations, but for the same muscle groups, intensity, volume, and duration. The position at the point of moderate discomfort will be self-adjusted by subjective perception over 12 weeks of intervention. The protocol model will change after seven weeks. In order to make the interventions more similar, the guide and videos of control group will be also sent to experimental group
  Arms: Active care group
Other: Active Comparator: Self-care group — The participants will receive counseling to stretching by guide and explanatory video that will be send by WhatsApp. The stretching exercise protocols will be the same performed by the experimental group. In addition, participants will receive recommendation to perform the protocol with the same weekly frequency, intensity, volume, and duration perform by the experimental group After the guide and explanatory video are sent, participants will receive a call for clarification. As well as in the experimental group, the protocol model will change after seven weeks; so, other guide and explanatory video will be sent for participants.
  Arms: Self-care group

SUMMARY:
This study is a randomized, single-blinded, parallel, superiority, controlled trial. The main objective is to verify the effects of a telehealth stretching exercise program on pain, depression, sleep parameters and functionality of women with fibromyalgia, during the Covid-19 pandemic. Participants will be women with primary fibromyalgia, seen at public and private health services, in the city of Pelotas (south of Brazil). Participants will be recruited through social networks, newspapers and support from the National Association of Fibromyalgia and Correlated Diseases (Anfibro). Eligible participants will be randomized, stratified by age (30 to 45; 46 to 60), and allocated to one of the two groups, experimental or control. The experimental group will receive a telehealth stretching exercise program twice a week (guided by a professional) and counseling guide to stretching exercises with explanatory video regarding the execution of the protocol proposed by the guide. The total duration of exercise program will be 40 minutes (will be 12 exercise, 3 sets of each stretching for 10 seconds, carried out individually by a video call application - WhatsApp). The control group will receive only counseling guide to stretching exercises with explanatory video regarding the execution of the protocol. Both interventions will last 12 weeks, with outcomes evaluations in three moments: baseline (week 0), midpoint (week 6) and after the intervention (week 13). The following outcomes will be evaluated: generalized index of pain, fatigue and severity of symptoms, depression, level of physical activity, functionality, quality of life and sleep. All outcomes will be evaluated by questionnaires self-completed, that will be answered on Google Docs by video call, with exception of functional test that will be applied by video call. The study's hypothesis consists of improving outcomes for both groups, but with superiority for the experimental group.

ELIGIBILITY:
Inclusion Criteria:

* Women between 30 and 60 years of age;
* Diagnosis of fibromyalgia (according medical confirmation) at least three months before eligibility;
* Inactive for at least three months;
* Inability or unwillingness to give informed consent for participation and to complete the questionnaires;
* Consent to participate in the study regardless of the allocation group.

Exclusion Criteria:

* Presence of another associated rheumatic pathology (secondary fibromyalgia);
* Uncontrolled systemic disease;
* Being under physiotherapeutic treatment;
* Lack of internet access.

Ages: 30 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Changes in the Widespread Pain Index | Zero week, six week, and twelve week
  A generalized pain index is a tool used to measure the amplitude of patients' clinical symptoms with fibromyalgia. It is considered a diagnostic scale, presenting 90.8% accuracy about the American College of Rheumatology's first criteria, de1990 and validated by the same institution in 2010 (WOLFE et al., 2010) being recognized by the Brazilian Society of Rheumatology - SBR, in 2017. Comprises the body areas usually affected by the disease, where the patient indicates if he felt pain at that moment in the last seven days (HEYMANN et al., 2017). Scores considered high are higher than 7. It will be checked if there was a change in painful behavior through collections in three periods of time, which will be compared at the end of the treatment.
Changes in Sleep Quality | Zero week, six week, and twelve week
  The Pittsburgh Sleep Quality Index Self-Report Questionnaire has been widely used to record sleep for four weeks. It includes 19 self-reported questions, divided into seven domains (HERNÁNDEZ et al., 2020) and five questions to be answered by the roommate, with questions about the noise produced during sleep. The score ranges from 0 to 3, where higher scores indicate worse sleep quality (BERTOLAZI et al., 2011). It was developed in 1989 by Buysse et al. and validated in the Brazilian version in 2011 by Bertolazi et al. (PASSOS et al., 2017). It is hoped to find a change in sleep quality; thus, three collections will be made, at different times of time, which will be compared at the end of the treatment.

SECONDARY OUTCOMES:
Symptom Severity Scale | Zero week, six week, and twelve week
  Symptom Severity, based on analyzing the primary symptoms reported in fibromyalgia, such as fatigue, sleep, and cognition, is considered a diagnostic criterion, with a sensitivity of 90.9% and specificity of 85.9% (HEYMANN et al., 2017). It comprises four domains, with scores ranging from 0 to 3, and scores above five are considered relevant. Validated by the American College of Rheumatology in 2010 (WOLFE et al., 2010) and recognized by the Brazilian Society of Rheumatology - SBR, 2017.
Impact of fibromyalgia on daily activities | Zero week, six week, and twelve week
  Fibromyalgia Impact Questionnaire (FIQ) is a survey that looks at the severity of the pathology on the individual's functional capacity and the perception of the quality of life. Their scores range from 0 to 100, where higher values indicate a more significant disease impact. Scores are expressed as follows: from 0 to 38 mild effect, from 39 to 58 moderate effect, and from 59 to 100 severe impact (UMAY et al., 2019) and validated in 1991 by Burckhardt et al., Translated and adapted for the Brazilian version in 2006, by Marques et al. (MARQUES et al., 2006).
Depressive symptoms | Zero week, six week, and twelve week
  Beck's Depression Inventory (BDI) is a tool whose purpose is to analyze the perception of depressive symptoms, developed and revised in 1996 by Becket al., And validated in the Brazilian version in 2012, by Gomes-Oliveira et al. (GOMES- OLIVEIRA et al., 2012). It includes 21 items, with scores ranging from 0 to 3, where the maximum score is 63, indicating severity. Values between 0 and 13 show minimal symptoms, 14 to 19 medium symptoms, 20 to 28 moderate, and 29 or more indicate severe depression (ALVENTOSA et al., 2020). Among the issues investigated there are feelings of sadness, failure, dissatisfaction, pessimism, self-judgment, distorted body vision, tiredness, lack of appetite, constant concerns, difficulty in work activities, and loss of libido (ANDRADE et al., 2020).
Physical activity level | Zero week, six week, and twelve week
  The participants' physical activity levels will be measured using the International Physical Activity Questionnaire - IPAQ-C, in its short version, including eight self-administered questions, in different domains such as work, leisure, domestic activities, and physical exercise. The data expressed in minutes, with the metabolic equivalent calculated (1 MET: 3.5 ml/kg/min). As with other questionnaires, we will apply it in electronic format, already tested and proven by previous studies (PIRES et al., 2014). Proposed and validated by the World Health Organization in 1998, it had its Brazilian version in 2001, through the study by Pardini et al. (PARDINIA et al., 2001).
Functionality / Flexibility | Zero week, six week, and twelve week
  Flexiteste is a tool developed by Araújo and Pavel in 1986 to analyze the flexibility of twenty articular movements of the human body (SALVADOR et al., 2010). Passively performed, with the examiner's aid up to the maximum joint amplitude, will adapt it for the online format, done in an active-assisted way, where the examined person assists the top angle, with the help of the opposite upper limb, with scores from 0 to 4. Higher values indicate increased mobility (ARAÚJO, 1986). The investigator masked will guide the patient's position remotely throughout the test.
Painful intensity at rest and movement | Zero week, six week, and twelve week
  Pain intensity will be analyzed using the Visual Analog Pain Scale - VAS, which comprises values from 0 to 10, where 0 corresponds to "no pain" and 10 "means the greatest pain imaginable" (HERNÁNDEZ et al., 2019). Being a unidirectional scale allows measuring the pain felt at the test's exact moment (MARTINEZ et al., 2011). The project will be used to check the pain at rest and right after the execution of a movement, aiming to understand the pain behavior before the proposed activity, in three moments: week 0, week six, and week 13. The associated test will elevate the upper limbs, with the hands splayed upwards and the fingers intertwined, using three sustained series of ten seconds, to be performed, together with the examiner's online presence. The EVA will be shown to the participant before the exercise and immediately after.
Subjective perception of well-being | Twelve week
  Will analyze the subjective perception of well-being through a simple question, "in your opinion, how much did participation in the project improve your feeling of general well-being," with structured responses based on the 5-point Likert Scale, varying from "dissatisfied" to "very satisfied." The same will be applied to the two groups in the same format as the questionnaires previously mentioned, through Google Docs, with a link to be made available on a scheduled date and time, through the WhatsApp application.

CONTACTS AND LOCATIONS:
Overall Officials: Cristine L Alberton, PhD, Principal Investigator — Federal University of Pelotas
Locations (1):
- Escola Superior de Educação Física, Pelotas, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Therapeutic physical exercise and supplements to treat fibromyalgia. — http://doi.org/10.1016/j.apunts.2017.07.001
- See also: Controlled, cross-sectional, multi-center study of physical capacity and associated factors in women with fibromyalgia — http://doi.org/10.1186/s12891-018-2047-1
- See also: Effectiveness of exercise on fatigue and sleep quality in fibromyalgia: a systematic review and meta-analysis of randomised trials. — http://doi.org/10.1016/j.apmr.2020.06.019
- See also: The efficacy of adding group behavioral activation to usual care in patients with fibromyalgia and major depression: design and protocol for a randomized clinical trial. — http://doi.org/10.1186/s13063-018-3037-1
- See also: Progress towards improved non-pharmacological management of fibromyalgia. — http://doi.org/10.1016/j.jbspin.2020.02.005
- See also: What happens to muscles in fibromyalgia syndrome — http://doi.org/10.1007/s11845-019-02138-w